CLINICAL TRIAL: NCT05841056
Title: Short Term Anti-aRrhythmic Therapy for Post-Operative AF in Cardiac Surgery Patients (START-POAF) Pilot Trial
Brief Title: Short Term Anti-aRrhythmic Therapy for Post-Operative AF in Cardiac Surgery Patients Pilot Trial
Acronym: START-POAF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.START-POAF
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation New Onset
Keywords: cardiac surgery; heart rhythm monitoring; amiodarone
MeSH Terms: interventions — Amiodarone

STUDY DESIGN:
Intervention Model Description: 1:1 ratio to receive amiodarone 200 mg maintenance therapy daily for four weeks or no maintenance therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amiodarone maintenance therapy (Active Comparator): Amiodarone 200 mg daily for four weeks
  Interventions: Drug: Amiodarone Hydrochloride 200 MG
- No Amiodarone maintenance therapy (No Intervention): No ongoing Amiodarone maintenance therapy for four weeks

INTERVENTIONS:
Drug: Amiodarone Hydrochloride 200 MG — 200 mg daily for 4 weeks
  Other Names: Pacerone; Cordarone
  Arms: Amiodarone maintenance therapy

SUMMARY:
The START-POAF pilot study is a prospective, open-label two-arm, randomized controlled trial with blinded assessment of outcomes (PROBE). This pilot study will assess Atrial Fibrillation (AF) recurrence and burden in patients with new-onset AF following cardiac surgery.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common abnormal heart rhythm in the world. In patients who have cardiac surgery, new AF is found as an early complication in more than one out of every four surgeries. In the weeks and months after heart surgery, patients who have new AF take a medication called amiodarone to keep their heart in rhythm as it heals. If the heart goes back into AF, patients can have symptoms of heart racing, heart failure (fluid on the lungs) or stroke. Although amiodarone is effective, it can have side effects like dizziness, nausea and slow heart rate. It may also damage the lungs, liver and thyroid gland. Many patients are not able to complete their full prescribed course after surgery. Therefore, it is crucial that the investigators find the shortest possible length of treatment with amiodarone that will keep the heart in rhythm while minimizing the chance of side effects or organ damage. The START-POAF Pilot Randomized Trial will compare two different durations of amiodarone treatment: 1) in-hospital load only and 2) in-hospital load plus 4 weeks after loading dose. All participants will wear an electrocardiogram (ECG) monitor for 4 weeks the day after they complete their loading dose. The investigators will compare the amount of AF seen on the ECG between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Have undergone cardiac surgery including CABG, valve surgery, ascending aorta replacement, or combinations thereof within 14 days of randomization;
3. Had new-onset POAF (or flutter), documented by 12-lead ECG or lasting ≥ 1 hour on telemetry. Patients can be in AF or sinus rhythm at the time of randomization;
4. Expected to receive 3 g - 5 g of amiodarone loading dose post-surgery.
5. Expected to be ready for hospital discharge within 48 h of randomization.

Exclusion Criteria:

1. Documented preoperative history of paroxysmal, persistent or permanent AF;
2. Planned use of a class I or III anti-arrhythmic drug (other than study drug);
3. Patients who have undergone heart transplant, complex congenital heart surgery, isolated ventricular assist device insertion, or AF ablation (surgical or catheter);
4. Known allergy to ECG adhesives;
5. Contraindication to amiodarone (i.e. hyperthyroidism, severe restrictive or obstructive lung disease, Long QT syndrome, PR > 240 ms, high-grade AV block).
6. Individuals who are pregnant, breastfeeding, or of childbearing potential - female subjects, premenopausal who are not surgically sterile, or, if sexually active not practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and, for those of childbearing potential, who have a positive pregnancy test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
3 patients per center per month | 2 years
  Ability to recruit an average of 3 participants per center per month
Less than 10% cross-over rate | 28 days
  Less than 10% cross-over rate
Intervention group taking at least 80% of their amiodarone 4 week maintenance therapy | 28 days
  Greater than and equal to 90% of the intervention group taking at least 80% of their amiodarone 4 week maintenance therapy
90% follow-up at 30 days | At 30 days post randomization date
  Greater than and equal to 90% follow-up at 30 days

SECONDARY OUTCOMES:
Burden of atrial fibrillation | In the 28 days measured by the continuous ECG monitor placed on the day after the participant finishes their 3-5g amiodarone loading dose
  Defined as percent time in atrial fibrillation
Time to first AF > 6 minutes, >6 hours and >24 hours | In the 28 days measured by the continuous ECG monitor placed on the day after the participant finishes their 3-5g amiodarone loading dose
  Time to first AF > 6 minutes, >6 hours and >24 hours reported from the continuous ECG monitor
Participants with at least one episode >6 minutes, >6 hours and >24 hours | In the 28 days measured by the continuous ECG monitor placed on the day after the participant finishes their 3-5g amiodarone loading dose
  Proportion of participants with at least one episode > 6 minutes, >6 hours and >24 hours reported from the continuous ECG

OTHER OUTCOMES:
Heart Failure | 90 days after randomization
  Number of participants who experience heart failure
Atrial Fibrillation | 90 days after randomization
  Number of participants who experience atrial fibrillation
A composite of stroke, myocardial infarction and cardiovascular death | 90 days after randomization
  Number of participants who have at least one of the following: stroke, myocardial infarction or cardiovascular death
Major bleeding | 90 days after randomization
  Number of participants who experience a major bleed
Systemic arterial embolism | 90 days after randomization
  Number of participants who experience a systemic arterial embolism
Atrial Fibrillation Effect on QualiTy of life (AFEQT) Questionnaire | Collected at baseline, 30 day follow-up and 90 day follow-up
  The Atrial Fibrillation Effect on Quality-of-life Questionnaire (AFEQT) evaluates symptoms, daily activities, and treatment concerns participants have related to atrial fibrillation and will be completed on all participants
SF-12 Questionnaire | Collected at baseline, 30 day follow-up and 90 day follow-up
  The SF-12 questionnaire which assesses physical and mental health will be completed on all participants
Electrical cardioversion | Randomization to 90 days
  Proportion of participants who undergo electrical cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: William McIntyre, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No